CLINICAL TRIAL: NCT01850160
Title: Efficacy and Safety of the Fixed-dose Combination of Valsartan Plus Chlorthalidone Vs Valsartan or Chlorthalidone Alone in the Treatment of Arterial Hypertension, Open-label, Controlled, Randomized and Multicenter Trial
Brief Title: Efficacy/Safety Study of Valsartan and Chlorthalidone Conjugate Treatment Compared to Simple Treatment for Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Farma de Colombia SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005-12 HTA
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Hypertension; High blood pressure; Drug therapy combination; Valsartan; Chlorthalidone; Safety; Efficacy
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Antihypertensive Agents; Angiotensin Receptor Antagonists; Sodium Chloride Symporter Inhibitors; Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GROUP A: Valsartan plus Chlorthalidone (Experimental): GROUP A: Combination therapy of Valsartan plus Chlorthalidone. Valsartan 80 mg/Chlorthalidone 12,5 mg. Once daily during 12 weeks.
  Interventions: Drug: GROUP A: Valsartan plus Chlorthalidone
- GROUP B: Valsartan (Experimental): GROUP B: Treatment with Monotherapy. Valsartan 80 mg. Once daily during 12 weeks.
  Interventions: Drug: GROUP B: Valsartan
- GROUP C: Chlorthalidone (Experimental): GROUP C: Treatment with Monotherapy. Chlorthalidone 12,5 mg. Once daily during 12 weeks.
  Interventions: Drug: GROUP C: Chlorthalidone

INTERVENTIONS:
Drug: GROUP A: Valsartan plus Chlorthalidone — Combination therapy of Valsartan plus Chlorthalidone: Valsartan 80 mg / Chlorthalidone 12,5 mg. Once daily during 12 weeks. If the goals of blood Pressure are uncontrolled at week 6, the dose will be increase to Valsartan 160 mg / Chlorthalidone 25 mg once daily.
  Other Names: Chlorthalidone Drug Combination; Valsartan Drug Combination; Antihypertensive Agents
  Arms: GROUP A: Valsartan plus Chlorthalidone
Drug: GROUP B: Valsartan — GROUP B: Treatment monotherapy: Valsartan 80 mg once daily during 12 weeks. If the goals of blood Pressure are uncontrolled at week 6, the dose will be increase to Valsartan 160 mg once daily.
  Other Names: Angiotensin II Receptor Antagonist; Antihypertensive Agents
  Arms: GROUP B: Valsartan
Drug: GROUP C: Chlorthalidone — GROUP C: Treatment monotherapy: Chlorthalidone 12,5 mg once daily during 12 weeks. If the goals of blood pressure are uncontrolled at week 6, the dose will be increase to Chlorthalidone 25 mg once daily.
  Other Names: Sodium Chloride Symporter Inhibitors; Antihypertensive Agents; Diuretics
  Arms: GROUP C: Chlorthalidone

SUMMARY:
This trial is aimed to assess the efficacy and safety of a fixed-dose combination therapy with Valsartan and Chlorthalidone, Vs Valsartan or Chlorthalidone alone for treatment of adult patients with diagnosis of arterial hypertension.

DETAILED DESCRIPTION:
In spite of the existence of a great variety of treatments with drugs effective against arterial hypertension, the percentages of arterial hypertension control with monotherapy remain quite low reason why the fixed-dose combinations of drugs have been one of the most interesting research topics in order to achieve an appropriate control of arterial hypertension.

The possibility of achieving better coverage and Blood Pressure control through a drug combination has leaded, on a scientific base of the efficacy of an Angiotensin Receptor Blockers II plus diuretic combination, to the development of a great number of combinations with different Angiotensin II Receptor Blockers plus hydrochlorothiazide. Yet it is noteworthy that despite the increasing evidence showing additional benefits in Blood pressure control and reduction of cardiovascular outcomes with chlorthalidone over hydrochlorothiazide, there is neither a great number of combinations nor studies with Angiotensin II Receptor Blockers plus chlorthalidone whereby the conduction of a trial assessing the efficacy and safety of Valsartan plus chlorthalidone in hypertensive patients is proposed plus the benefits of combination therapy that include, among others, the greater efficacy with lower doses of each individual component as well as reduction in occurrence of adverse events directly related with lower drug doses.With this treatment schedule it is expected to obtain higher control of blood pressure values and greater percentage of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of arterial hypertension defined as:
* Systolic blood pressure greater or equal to 140 and lower than 180 mmHg
* Diastolic blood pressure greater or equal to 90 and lower than 110 mmHg
* Non controlled patients with antihypertensive treatment (blood pressure values: Systolic blood pressure > 140 mmHg and/or Diastolic blood pressure > 90 mmHg) or patients antihypertensive treatment-naïve.
* Likelihood of attending consultations according to the trial chronogram.
* Informed Consent Signature.

Exclusion Criteria:

* Diagnosis of severe or malignant arterial hypertension defined as:
* Systolic blood pressure greater or equal to 180 mmHg
* Diastolic blood pressure greater or equal to 110 mmHg
* Patients with secondary arterial hypertension of any etiology.
* Pregnant women or women with childbearing potential who are not using appropriate contraception methods; women planning to become pregnant during the trial.
* Patients with history of Acute Myocardial Infarction o Angina Pectoris within the 6 months prior to the trial initiation.
* Diagnosis of Cerebrovascular Disease (CVD) o Transient Ischemic Attack (TIA) within the 6 previous months.
* Patients with Severe Renal Disease defined by serum Creatinine levels higher than 1.5 mg/dl.
* Diagnosed or suspected unilateral or bilateral renal artery stenosis.
* History of non remitting cancer within the 5 years prior to the trial initiation.
* Patients with Hypokalemia or Hyperkalemia.
* Patients receiving Valsartan or Chlortalidone during the 14 previous days.
* Patients with known hypersensitivity to Valsartan or Chlorthalidone.
* Unstable patients with antecedent of hospitalization within the 4 days prior to their enrollment in the trial.
* Patients with history of drugs and alcohol abuse within the last year.
* Patients who have taken part in other clinical trial within the 4 weeks prior to the initiation of this research.
* Patients with any other clinical condition that the investigator deems may affect the patient follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of the fixed-dose combination treatment with Valsartan plus Chlorthalidone | 12 weeks
  Efficacy and safety of a fixed-dose combination treatment of Valsartan plus Chlorthalidone Vs Valsartan or Chlorthalidone alone in the treatment of patients with arterial hypertension

SECONDARY OUTCOMES:
Changes in Systolic and Diastolic Blood pressure values | 12 weeks
  Assess the changes in Systolic and Diastolic Blood Pressure from baseline up to week 12
Changes of Systolic blood pressure values | 12 weeks
  Assess the changes of systolic blood pressure from baseline up to week 6 and 12
Changes of Diastolic blood pressure values | 12 weeks
  Assess the changes of diastolic blood pressure from baseline up to week 6 and 12
Changes of diastolic blood pressure in arterial blood pressure median values | 12 weeks
  Assess the changes in diastolic blood pressure in Arterial Blood Pressure Media from baseline up to week 12
Changes of systolic blood pressure values in arterial blood pressure median values | 12 weeks
  Assess the change in systolic blood pressure in Arterial Blood Pressure Median from baseline up to week 12
Patient that achieving blood pressure values lower than 140/90 (systolic/diastolic) at week 6 and 12 | 12 weeks
  Determine the percentage of patients achieving blood pressure values lower than 140/90 (systolic/diastolic) at weeks 6 and 12
Patients that achieving systolic blood pressure values lower than 140 at week 6 and 12 | 12 weeks
  Determine the percentage of patients achieving systolic blood pressure lower than 140 at weeks 6 and 12
Patients that achieving diastolic blood pressure values lower than 90 at week 6 and 12 | 12 weeks
  Determine the percentage of patients achieving diastolic blood pressure lower than 90 at week 6 and 12

OTHER OUTCOMES:
Metabolic changes secondary to the treatment with Valsartan and Chlorthalidone, Vs Valsartan or Chlorthalidone | 12 weeks
  Identify if there are significant differences regarding metabolic changes secondary to the treatment with Valsartan and Chlorthalidone Vs Valsartan or Chlorthalidone.
Incidence of adverse events in each intervention group | 12 weeks
  Determine the percentage of incidence of adverse events in each intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Romero, MD, Study Director — Farma de Colombia SA
Locations (8):
- Colombia (3):
  - MedPlus, Bogota DC, Bogota DC
  - Centro de Diagnostico Cardiologico, Cartagena, Departamento de Bolívar
  - Fundacion Cardiomet Cequin, Armenia, Quindío Department
- Ecuador (5):
  - Centro AMCOR, Quito
  - Centro Clinico quirurgico, Quito
  - Centro médico de hipertensión arterial, Quito
  - Clínica DAME, Quito
  - Consultorio Edificio Novoa, Quito

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manzur F, Rico A, Romero JD, Rodriguez-Martinez CE. Efficacy and Safety of Valsartan or Chlorthalidone vs. Combined Valsartan and Chlorthalidone in Patients With Mild to Moderate Hypertension: The VACLOR Study. Clin Med Insights Cardiol. 2018 Sep 3;12:1179546818796482. doi: 10.1177/1179546818796482. eCollection 2018. PMID 30202211